CLINICAL TRIAL: NCT06338371
Title: The Effect of Pelvic Floor Muscle Exercise on Sexual Function in Women of Reproductive Age:A Randomized-Controlled Tria
Brief Title: Effect of Pelvic Floor Muscle Exercise on Sexual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serap Tekbas (Other)
Responsible Party: Sponsor-Investigator, Serap Tekbas, Principal Investigator, Izmir Tinaztepe University
Organization: Izmir Tinaztepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IZTU-TEKBAŞ-001
Record Dates: First submitted 2024-03-17; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Floor Muscle Weakness; Sexuality
Keywords: Pelvic floor muscle; exercise; sexual function; reproductive age
MeSH Terms: conditions — Sexuality; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Content (Experimental): Group receiving training on pelvic floor exercise
  Interventions: Behavioral: Pelvic Floor exercise training
- Control Group (No Intervention): Untrained group

INTERVENTIONS:
Behavioral: Pelvic Floor exercise training — The level of sexual function was determined by implementing FSFI for all individuals included in the sample. The participants were divided into two groups, control and training groups, using the randomization program on the computer. Pelvic floor exercise training was given to one group. Trainings were conducted online on different days. Each training lasted 120 minutes. After training was completed, women in the training group were instructed to perform three sets of 8-12 repetitive pelvic floor muscle contractions per day and to use an exercise diary to record their practice. Women in the training group were also given a booklet and the recording of the training video was shared. the training, a brochure explaining how to perform the pelvic floor muscle exercises, which was included in the training content, was prepared and delivered to the training group on the first day of each week. After the training, FSFI was applied to both groups 3 times, in the 1st, 2nd, and 3rd months.
  Arms: Training Content

SUMMARY:
The goal of this evaluate the effect of pelvic floor muscle exercises on sexual function in women of reproductive age. A randomized controlled trial was conducted in a sample of women of reproductive age, 77 women were randomly assigned to control (n=39) and training (n=38) groups. A form including questions regarding socio-demographic characteristics and the Female Sexual Function Index was applied to all women included in the study. Pelvic floor exercise training was given to the women in the training group and the Female Sexual Function Index was applied to both groups in the 1st, 2nd, and 3rd months. The differences between those who received and those who did not receive training and the effects of regular pelvic exercise on sexual function were evaluated by month.

Research Hypotheses H1: Sexual function scores of women of reproductive age who regularly perform pelvic floor muscle exercises are higher than those who do not exercise.

H2: Sexual function scores are higher for those who regularly exercise their pelvic floor muscles for at least two months

DETAILED DESCRIPTION:
The research has a prospective, randomized controlled design.

Inclusion criteria of the study:

Women aged between 18-49 who agreed to participate in the study and who had a regular sexual life were included in the study.

Exclusion criteria of the study:

Women who did not have a regular sex life, who had undergone an operation that prevented them from doing pelvic floor exercises, and who exercised regularly because it could strengthen the pelvic muscles and affect the results of the study were excluded from the study. In addition, menopausal women were not included in the study

The purpose of the research was explained and women between the ages of 18-49 were invited to participate from social media platforms. The level of sexual function was determined by implementing FSFI for all individuals included in the sample. The participants were divided into two groups, control and training groups, using the randomization program on the computer. Pelvic floor exercise training was given to one group. The training was given online due to the COVID-19 pandemic. Four groups were formed for the training. Three groups consisted of ten people and one group of eight people. Trainings were conducted online on different days. Each training lasted 120 minutes. 70 minutes of the training consisted of theoretical information, 30 minutes of the training consisted of watching videos about the application of pelvic floor exercises, and the last 20 minutes consisted of taking the questions of the participants on the subject and answering these questions. After training was completed, women in the training group were instructed to perform three sets of 8-12 repetitive pelvic floor muscle contractions per day and to use an exercise diary to record their practice. Women in the training group were also given a booklet and the recording of the training video was shared. the training, a brochure explaining how to perform the pelvic floor muscle exercises, which was included in the training content, was prepared and delivered to the training group on the first day of each week. After the training, FSFI was applied to both groups (who received and did not receive the training) 3 times, in the 1st, 2nd, and 3rd months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-49
* Women who have not entered menopause
* Women with regular sexual life.

Exclusion Criteria:

* Women in menopause
* Women diagnosed with gynecological cancer
* Women who do not have a regular sexual life

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A study was planned in which the sample group consisted only of women.
Enrollment: 77 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Determining Number of Participants | Baseline (Before training)
  Power calculation was made to determine the size of the sample constituting the training and control groups. In the power analysis performed for the training and control groups in line with the literature data [(SD±6.5) with an α of 5% and a power of 80% (1-ß)], the expected sample size was determined as a total of 68 people, 34 in the training group and 34 in the control group13. However, considering the possible data loss, it was decided to include 40 individuals in each group. Data were collected using Google Forms through social media platforms. Women who volunteered to participate in the study were invited and written consent was taken from the individuals included in the study. 80 women who agreed to participate were included in the study of women who agreed to participate in the study. Sample group n=80
Initial scale application | Baseline (Before training)
  Women's Descriptive Characteristics: The form was prepared by the researcher in line with the literature and consists of 23 questions regarding sociodemographic characteristics, general health status, and obstetric characteristics of women.
  Female Sexual Function Index (FSFI): The scale was created by Rosen et al. in 2000 in order to evaluate sexual function. It includes 19 questions and evaluates desire, arousal, lubrication, orgasm, satisfaction, and pain in a multidimensional way. The highest raw score obtainable from the index is 36 and the lowest raw score is 2. An increase in the scores on the total index and the sexual desire, arousal, lubrication, orgasm, and general satisfaction subscales indicate an improvement in all these parameters.
Distribution of participants into groups | Baseline (Before training)
  The sample group was randomly divided into training and control. The study protocol for the trial was created using SPIRIT guidelines and the trial reporting was created according to the CONSORT checklist. In order to avoid selection bias in the study, patients were assigned to the experimental and control groups with the block randomization method. The n=80 samples included in the study were randomly divided into case (n=40) and control (n=40) groups with the help of the "Random Allocation Software" computer program.

SECONDARY OUTCOMES:
Providing pelvic floor exercise for training group | Baseline (Before training)
  Pelvic Floor Muscle Exercise training was given implemented to the training group Pelvic floor exercise training was given to the control group. A 120-minute training program was created to implement pelvic floor muscle exercises and explain the pelvic muscles. 70 minutes of the training consisted of theoretical information, 30 minutes of watching videos on the application of pelvic floor exercises, and the last 20 minutes of the training consisted of taking and answering questions from the participants on the subject.
Female Sexual Function Index | 1st Month
  Female Sexual Function Index (FSFI): The scale was created by Rosen et al. in 2000 in order to evaluate sexual function. It includes 19 questions and evaluates desire, arousal, lubrication, orgasm, satisfaction, and pain in a multidimensional way. The highest raw score obtainable from the index is 36 and the lowest raw score is 2. An increase in the scores on the total index and the sexual desire, arousal, lubrication, orgasm, and general satisfaction subscales indicate an improvement in all these parameters.
Female Sexual Function Index | 2st Month
  Female Sexual Function Index (FSFI): The scale was created by Rosen et al. in 2000 in order to evaluate sexual function. It includes 19 questions and evaluates desire, arousal, lubrication, orgasm, satisfaction, and pain in a multidimensional way. The highest raw score obtainable from the index is 36 and the lowest raw score is 2. An increase in the scores on the total index and the sexual desire, arousal, lubrication, orgasm, and general satisfaction subscales indicate an improvement in all these parameters.
Female Sexual Function Index | 3st Month
  Female Sexual Function Index (FSFI): The scale was created by Rosen et al. in 2000 in order to evaluate sexual function. It includes 19 questions and evaluates desire, arousal, lubrication, orgasm, satisfaction, and pain in a multidimensional way. The highest raw score obtainable from the index is 36 and the lowest raw score is 2. An increase in the scores on the total index and the sexual desire, arousal, lubrication, orgasm, and general satisfaction subscales indicate an improvement in all these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Tekbaş, Principal Investigator — Head of Midwifery Department
Locations (1):
- Izmir Tinaztepe University, Izmir, Buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eftekhar T, Dashti M, Shariat M, Haghollahi F, Raisi F, Ghahghaei-Nezamabadi A. Female Sexual Function During the Menopausal Transition in a Group of Iranian Women. J Family Reprod Health. 2016 Jun;10(2):52-8. PMID 27648093
- [Derived] Tekbas S. The effect of pelvic floor muscle exercise on sexual function in women of reproductive age: A randomized controlled trial. Medicine (Baltimore). 2025 Sep 12;104(37):e44324. doi: 10.1097/MD.0000000000044324. PMID 40958332
- See also: DeUgarte CM, Berman L, Berman J. Female sexual dysfunction-from diagnosis to treatment. Sexuality, Reproduction and Menopause 2004; 2 (3), 139-145. — http://doi.org/10.1016/j.sram.2004.07.002
- See also: Wright JJ, O'Connor KM. Female sexual dysfunction. Medical Clinics of North America 2015; 99 (3), 607-628 — http://doi.org/10.1016/j.mcna.2015.01.011
- See also: Kanter G, Rogers RG, Pauls RN, Kammerer-Doak, D, Thakar, RA strong pelvic floor is associated with higher rates of sexual activity in women with pelvic floor disorders. International urogynecology journal 2015; 26(7), 991-996 — http://doi.org/10.1007/s00192-014-2583-7